CLINICAL TRIAL: NCT04231916
Title: High Resolution Thermal Imaging to Identify Vertebral Fractures in Children and Young People With Osteogenesis Imperfecta
Acronym: THERMOI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: SCH-13-067b
Record Dates: First submitted 2020-01-03; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta

ARMS (1):
- Patients aged 5-18 years (Experimental): Patients with Osteogenesis Imperfecta (with known vertebral fractures)for phase one of the study.
  Patients with Osteogenesis Imperfecta for phase 2 of the study In both groups patients will be aged 5 years and over
  Interventions: Device: Thermal imaging device

INTERVENTIONS:
Device: Thermal imaging device

SUMMARY:
Brittle bone disease also known as osteogenesis imperfecta (OI) is characterised by a defect in the bone tissue that leads to recurrent fractures and significant bone deformities in children. These fractures include vertebral (spinal) fractures. As a result, child with OI require regular clinic surveillance that includes repeated xrays of the spine. in our pilot study the investigators plan to use a thermal imaging camera that can pick up changes in temperature to 0.03 degrees to determine whether the investigators can accurately identify vertebral fractures without the need for radiation. in the first part of the study the investigators will compare the thermal images from the camera with the xrays to see if the investigators can pick up the vertebral fractures seen on the xray picture. If this is possible, then the investigators will move on to phase 2 of the study which will investigate the ability of the thermal camera to pick up vertebral fractures without prior knowledge of where the fractures are located. If this approach is successful this will help us to develop a nonradiation, lowcost painless way of identifying vertebral fractures in children with OI.

ELIGIBILITY:
* Patients with Osteogenesis Imperfecta (with known vertebral fractures)for phase one of the study.
* Patients with Osteogenesis Imperfecta for phase 2 of the study
* In both groups patients will be aged 5 years and over

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2016-07-07 (Actual); Study Completion 2016-07-07 (Actual)

PRIMARY OUTCOMES:
Thermal imaging device | 15 minutes
  The ability to pick up vertebral morphology and fractures in relation to spine X-rays